CLINICAL TRIAL: NCT01887964
Title: Dietary Fiber Intervention in Hutterite Population of South Dakota With and Without Signs of Metabolic Syndrome
Brief Title: Effect of Resistant Starch (Type-4) on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Moul Dey, Associate Professor, South Dakota State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1112012-CR
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Syndrome
Keywords: Diabetes; Obesity; Cardiovascular disease; Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-1 (Other): Received control flour first and then Resistant starch type 4 (RS4) flour
  Interventions: Other: RS4 enriched flour; Other: Control flour
- Community-2 (Other): Received RS4 flour first and then control flour
  Interventions: Other: RS4 enriched flour; Other: Control flour

INTERVENTIONS:
Other: RS4 enriched flour — Wheat flour with 30% resistant starch (type-4)
Other: Control flour — Wheat flour without resistant starch (type-4)

SUMMARY:
Metabolic syndrome is a condition characterized by excess body weight, large waist circumference, high cholesterol and glucose in the blood, and hypertension. People with metabolic syndrome are at increased risk for heart diseases. Research shows benefits of regular fiber intake in metabolic syndrome. However, due to altered taste and texture of the high fiber foods, long term intake of fiber is a challenge for metabolic syndrome patients. This study is designed to find if blinded-substitution of regular wheat flour in domestic kitchen with wheat flour enriched by an adaptable type of fiber (resistant starch-4), minimizes metabolic syndrome symptoms. this special type of fiber is also obtained from wheat.

ELIGIBILITY:
Inclusion Criteria:

- Any individual aged 18-80 years

Exclusion Criteria:

* Pregnant
* Lactating
* Requires special diets or dietary regimens
* On long term antibiotic therapy
* Diagnosed with gastrointestinal diseases (Irritable Bowel syndrome, Crohn's disease or Colitis)
* Immune compromised
* Have cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in metabolic syndrome risk components | 26 weeks

SECONDARY OUTCOMES:
Changes in anthropometric outcomes | 26 weeks
  Body weight, body mass index, systolic and diastolic blood pressure, fat mass and fat-free mass
Changes in blood lipid profile | 26 weeks
  total cholesterol, LDL cholesterol, HDL cholesterol, non-HDL cholesterol and triglycerides
Changes in blood glucose indices | 26 weeks
  fasting blood glucose, postprandial blood glucose and Hemoglobin-A1C

CONTACTS AND LOCATIONS:
Overall Officials: Moul Dey, PhD, Principal Investigator — South Dakota State University; Bonny Specker, PhD, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant's identity will not be shared. This clinical trial is complete. All results were published as two research articles: PMCID: PMC4928084 and PMCID: PMC4048643. Raw sequence data were submitted to Sequence Read archive as referenced in the manuscript PMC4928084.

REFERENCES:
- [Derived] Dhakal S, Dey M. Resistant starch type-4 intake alters circulating bile acids in human subjects. Front Nutr. 2022 Oct 20;9:930414. doi: 10.3389/fnut.2022.930414. eCollection 2022. PMID 36337613